CLINICAL TRIAL: NCT01880697
Title: A Phase III, Open-Label, Single-Arm, Multicenter Study to Evaluate the Safety and Immunogenicity of a Trivalent, Surface Antigen Inactivated Subunit Influenza Virus Vaccine Produced in Mammalian Cell Culture (Optaflu®) in Healthy Adults
Brief Title: Safety and Immunogenicity of a Cell Derived Subunit Trivalent Nonadjuvanted Influenza Study Vaccine in Adults Aged 18 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V58_33S; 2013-000621-30 (EudraCT Number)
Record Dates: First submitted 2013-06-12; First posted 2013-06-19 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2013-12

CONDITIONS: Human Influenza
Keywords: Influenza; adults; elderly; immunology; safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TIVc (≥18 to ≤ 60 years) + TIVc (≥ 61 years) (Experimental): Subjects in each age cohort received one dose of the cell-derived trivalent, surface antigen inactivated subunit influenza virus vaccine (TIVc) formulation 2013/2014 Northern Hemisphere
  Interventions: Biological: TIVc

INTERVENTIONS:
Biological: TIVc — Trivalent Influenza Virus Vaccine (surface antigen, inactivated, cell-based)

SUMMARY:
The present study is designed to confirm the safety and immunogenicity of cell-derived, trivalent, surface antigen, inactivated influenza vaccine in 2 age cohorts: 18 to ≤60 years and ≥61 years and the antibody response to each influenza vaccine antigen, as measured by Single Radial Hemolysis (SRH) or Hemagglutination Inhibition (HI) at approximately 21 days post immunization. The vaccine composition will be based on the WHO-recommended influenza strains for the 2013/2014 Northern Hemisphere vaccine. The results of this study are intended to support the use of this vaccine in future influenza seasons if the recommended vaccine composition remains the same, in compliance with the requirements of the current EU recommendations for clinical trials related to yearly licensing of influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteer ages 18 years or older, mentally competent, willing and able to give written informed consent prior to study entry;
* Able to comply with all the study requirements; and
* In good health as determined by the outcome of medical history, physical examination, and clinical judgment of the investigator

Exclusion Criteria:

* Had behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, might have interfered with the subject's ability to participate in the study;
* Had a serious chronic or acute disease (in the judgment of the investigator) including, but not limited to

  * medically significant cancer (except for benign or localized skin cancer, cancer in remission for ≥10 years, or localized prostate cancer that has been clinically stable for >2 years without treatment)
  * medically significant advanced congestive heart failure (ie, New York Heart Association [NYHA] class III and IV)
  * chronic obstructive pulmonary disease (ie, Global initiative for chronic Obstructive Lung Disease [GOLD] stage III and IV)
  * autoimmune disease (including rheumatoid arthritis and excepting Hashimoto's thyroiditis that has been clinically stable for ≥5 years)
  * diabetes mellitus type I
  * poorly controlled diabetes mellitus type II
  * advanced arteriosclerotic disease
  * history of underlying medical condition such as major congenital abnormalities requiring surgery, chronic treatment, or associated with developmental delay (Down's syndrome)
  * acute or progressive hepatic disease
  * acute or progressive renal disease
  * severe neurological (especially Guillain-Barré syndrome) or psychiatric disorder
  * severe asthma
* Had a history of any anaphylactic reaction and/or serious allergic reaction to any component of the study vaccine;
* Had a known or suspected (or had a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting, for example, from:

  * receipt of immunosuppressive therapy (any parenteral or oral corticosteroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study,
  * receipt of immunostimulants within the past 6 months,
  * receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivates within the past 3 months and for the full length of the study, or
  * suspected or known human immunodeficiency virus (HIV) infection or HIV-related disease
* Had known or suspected drug or alcohol abuse within the past 2 years;
* Had bleeding diathesis or conditions associated with prolonged bleeding time that, in the investigator's opinion, would have interfered with the safety of the subject;
* Was not able to comprehend and to follow all required study procedures for the whole period of the study;
* Had a history or any illness that, in the opinion of the investigator, would have posed additional risk to the subjects because of participation in the study;
* Had the following within the past 6 months:

  * had any laboratory-confirmed seasonal or pandemic influenza disease
  * received any seasonal or pandemic influenza vaccine
* Had received any other vaccine within 4 weeks prior to enrollment in this study or who were planning to receive any vaccine during the study;
* Had acute or chronic infections requiring antiviral therapy within the last 7 days;
* Had experienced fever (ie, body temperature [preferably oral] ≥38.0°C) within the last 3 days of intended study vaccination;
* Had participated in any clinical trial with another investigational product 4 weeks prior to first study visit or intended to participate in another clinical study at any time during the conduct of this study;
* Was part of study personnel or has close family members conducting this study;
* Had a body mass index (BMI) >35 kg/m2 (BMI is calculated by dividing the subject's weight in kilograms by the subject's height in meters multiplied by the subject's height in meters);
* Was pregnant (confirmed by positive urine pregnancy test) or nursing (breastfeeding) or was a female of childbearing potential who refused to use an acceptable method of birth control for the whole duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (1):
- Rostock University, Department of Tropical Medicine and Infectious Diseases, Ernst Heydemann Strasse 6, Rostock, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- TIVc (≥18 to ≤ 60 Years): Adult subjects received one dose of the cell-derived trivalent, surface antigen inactivated subunit influenza virus vaccine (TIVc) formulation 2013/2014 Northern Hemisphere
- TIVc (≥ 61 Years): Elderly subjects received one dose of the cell-derived trivalent, surface antigen inactivated subunit influenza virus vaccine (TIVc) formulation 2013/2014 Northern Hemisphere
Period: Overall Study
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years)
Started | 63 | 63
Completed | 63 | 62
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years) | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (10.7) | 68.3 (4.8) | 53.8 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 71
  Male | 25 | 30 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Single Radial Hemolysis (SRH) Areas ≥25mm2, Against Each of Three Vaccine Strains After Receiving One Dose of TIVc
Description: Immunogenicity was assessed in terms of percentages of subjects in both age groups with SRH areas ≥25mm2 against each of the three vaccine strains, three weeks after receiving one dose of TIVc.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if the percentage of subjects achieving post vaccination SRH areas ≥ 25mm2 is >70% for adults aged 18 to ≤60 years and >60% for subjects aged ≥61 years.
Time Frame: Day 22 (vaccination is on day 1)
Population: Analysis was done on the per-protocol population i.e all subjects who have received study vaccination and provided immunogenicity data both at baseline and after vaccination; did not withdraw informed consent and did not have RT-PCR confirmed influenza during the study.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years)
Number analyzed (Participants) | 62 | 61
Percentages of Subjects
  Day 1/baseline (H1N1 strain) | 66 [53 to 78] | 41 [29 to 54]
  Day 22 (H1N1 strain) | 98 [91 to 100] | 84 [72 to 92]
  Day 1/baseline (H3N2 strain) | 44 [31 to 57] | 39 [27 to 53]
  Day 22 (H3N2 strain) | 92 [82 to 97] | 77 [65 to 87]
  Day 1/baseline (B strain) | 68 [55 to 79] | 77 [65 to 87]
  Day 22 (B strain) | 98 [91 to 100] | 98 [91 to 100]

2. Primary Outcome: Percentages of Subjects With Seroconversion or Significant Increase in SRH Area, Against Each of Three Vaccine Strains After Receiving One Dose of TIVc
Description: Immunogenicity was assessed in terms of percentages of subjects in both age groups achieving seroconversion or significant increase by SRH area against each of the three vaccine strains ,three weeks after receiving one dose of TIVc.
  Seroconversion is defined as percentage of subjects with a pre-vaccination SRH area ≤4mm2 achieving a post-vaccination SRH area ≥25 mm2. Significant increase is defined as percentage of subjects with a pre-vaccination SRH area >4mm2 achieving at least 50% increase in post-vaccination SRH area.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if the percentage of subjects achieving post vaccination SRH areas ≥ 25mm2 is >40% for adults aged 18 to ≤60 years and >30% for subjects aged ≥61 years.
Time Frame: Day 22 (vaccination is on day 1)
Population: Analysis was done on the per-protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years)
Number analyzed (Participants) | 62 | 61
Percentages of Subjects
  H1N1 | 68 [55 to 79] | 56 [42 to 68]
  H3N2 | 65 [51 to 76] | 46 [33 to 59]
  B | 58 [45 to 70] | 39 [27 to 53]

3. Primary Outcome: Geometric Mean Ratio of Post Vaccination Versus Pre Vaccination Geometric Mean Areas (GMAs), After One Dose of TIVc
Description: The antibody responses were evaluated in terms of GMRs of post vaccination GMAs to pre vaccination GMAs against each of the three vaccine strains, three weeks after receiving one dose of TIVc The related European (CHMP) criterion for the assessment of immunogenicity is met if the GMR day 22/day 1 is >2.5 for adults aged 18 to ≤60 years and > 2.0 in for subjects aged ≥61 years.
Time Frame: Day 22/day 1
Population: Analysis was done on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years)
Number analyzed (Participants) | 62 | 61
Ratio
  H1N1 | 2.89 [2.16 to 3.86] | 3.14 [2.29 to 4.31]
  H3N2 | 2.52 [2.03 to 3.12] | 2.05 [1.67 to 2.53]
  B | 1.82 [1.54 to 2.16] | 1.5 [1.28 to 1.76]

4. Primary Outcome: Percentage of Subjects With Haemagglutination Inhibition (HI) Titers ≥40, Against Each of Three Vaccine Strains After Receiving One Dose of TIVc
Description: Immunogenicity was assessed in terms of percentages of subjects in both age groups with HI titers ≥40, against each of the three vaccine strains, three weeks after receiving one dose of TIVc.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if the percentage of subjects achieving HI titers ≥ 40 is >70% for adults aged 18 to ≤60 years and >60% for subjects aged ≥61 years.
Time Frame: Day 22 (vaccination is on day 1)
Population: Analysis was done on the per-protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years)
Number analyzed (Participants) | 62 | 61
Percentages of Subjects
  Day 1/baseline (H1N1 strain) | 68 [55 to 79] | 66 [52 to 77]
  Day 22 (H1N1 strain) | 100 [94 to 100] | 97 [89 to 100]
  Day 1/baseline (H3N2 strain) | 89 [78 to 95] | 87 [76 to 94]
  Day 22 (H3N2 strain) | 97 [89 to 100] | 95 [86 to 99]
  Day 1/baseline (B strain) | 58 [45 to 70] | 46 [33 to 59]
  Day 22 (B strain) | 94 [84 to 98] | 80 [68 to 89]

5. Primary Outcome: Percentages of Subjects With Seroconversion or Significant Increase in HI Antibody Titers After Receiving One Dose of TIVc
Description: Immunogenicity was assessed in terms of percentages of subjects in both age groups achieving seroconversion or significant increase in HI antibody titers after receiving one dose of TIVc.
  Seroconversion is defined as percentage of subjects with a pre-vaccination HI titer <10 to a post-vaccination titer ≥40. Significant increase is defined as percentage of subjects with a pre-vaccination HI titer >10 to at least a 4-fold increase in post-vaccination HI antibody titers.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if >40 % for adults aged 18 to ≤60 years and >30% for subjects aged ≥61 years achieve seroconversion or significant increase in post-vaccination HI titers.
Time Frame: Day 22 (vaccination is on day 1)
Population: Analysis was done on the per-protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years)
Number analyzed (Participants) | 62 | 61
Percentages of Subjects
  H1N1 | 63 [50 to 75] | 43 [30 to 56]
  H3N2 | 47 [34 to 60] | 26 [16 to 39]
  B | 48 [35 to 61] | 28 [17 to 41]

6. Primary Outcome: Geometric Mean Ratio of Post Vaccination Versus Pre Vaccination HI Antibody Titers, Against Each of Three Vaccine Strains After Receiving One Dose of TIVc
Description: The antibody responses following one dose of TIVc were evaluated in terms of GMRs of post vaccination against pre vaccination geometric mean HI titers against each of the three vaccine strains, three weeks after receiving one dose of TIVc.
  The related European (CHMP) criterion for the assessment of immunogenicity is met if the GMR day 22/day 1 is >2.5 for adults aged 18 to ≤60 years and > 2.0 for subjects aged ≥61 years.
Time Frame: Day 22/day 1
Population: Analysis was done on the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years)
Number analyzed (Participants) | 62 | 61
Ratio
  H1N1 | 8.8 [5.66 to 14] | 3.61 [2.61 to 5.01]
  H3N2 | 3.52 [2.4 to 5.15] | 2.22 [1.63 to 3.01]
  B | 3.31 [2.45 to 4.47] | 2.4 [1.81 to 3.17]

7. Primary Outcome: Number of Subjects Reporting Solicited Adverse Events After Receiving One Dose of TIVc
Description: The number of adult and elderly subjects reporting solicited local and systemic adverse events and other solicited adverse events after receiving one dose of TIVc are reported.
Time Frame: Day 1 to Day 4 post-vaccination
Population: Analysis was done on the solicited safety set population i.e all subjects who have post-vaccination AE or reactogenicity records.
Measure: Number; unit: Subjects
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years)
Number analyzed (Participants) | 63 | 63
Subjects
  Any local | 32 | 18
  Injection site induration | 5 | 1
  Injection site erythema | 1 | 1
  Injection site ecchymosis | 1 | 0
  Injection site pain | 31 | 18
  Any systemic | 17 | 8
  Chills/shivering | 1 | 1
  Malaise | 3 | 2
  Myalgia | 1 | 1
  Arthralgia | 3 | 3
  Headache | 11 | 6
  Fatigue | 10 | 2
  Fever | 1 | 0
  Prophylactic use of analgesics/antipyretics | 2 | 0
  Therapeutic use of analgesics/antipyretics | 2 | 1

8. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Receiving One Dose of TIVc
Description: The number of subjects in both age groups reporting any unsolicited AEs (between Day 1 to 4), serious adverse events (SAEs), medically attended AEs, AEs leading to premature withdrawal (throughout the study period), after receiving one dose of TIVc is reported.
Time Frame: Day 1 through Day 22 post-vaccination
Population: Analysis was done on the unsolicited safety set population i.e all subjects who have post-vaccination AE or reactogenicity records.
Measure: Number; unit: Subjects
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years)
Number analyzed (Participants) | 63 | 63
Subjects
  Any AEs | 6 | 4
  At least possibly related AEs | 2 | 0
  Serious AEs | 1 | 0
  At least possibly related SAEs | 0 | 0
  Medically attended AEs | 4 | 3
  AEs leading to discontinuation | 0 | 0
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: All solicited AEs and unsolicited AEs collected from Day 1 to Day 4; serious adverse events (SAEs), medically attended AEs, AEs leading to premature withdrawal collected from Day 1 to Day 22.
Arm/Group | TIVc (≥18 to ≤ 60 Years) | TIVc (≥ 61 Years)
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/63
Other Adverse Events (participants affected / at risk) | 36/63 | 22/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIVc (≥18 to ≤ 60 Years) (N=63) | TIVc (≥ 61 Years) (N=63)
Tooth infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIVc (≥18 to ≤ 60 Years) (N=63) | TIVc (≥ 61 Years) (N=63)
Headache (Nervous system disorders) | 11 | 6
Fatigue (General disorders) | 10 | 2
Injection site induration (General disorders) | 4 | 1
Injection site pain (General disorders) | 32 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days